CLINICAL TRIAL: NCT05341869
Title: PREEMPTİVE PARA-CERVİCAL BLOCK FOR POSTOPERATİVE PAIN AFTER LAPAROSCOPIC HYSTERECTOMY: A RANDOMIZED PLACEBO CONTROLLED TRIAL
Brief Title: PREEMPTİVE PARA-CERVİCAL BLOCK FOR POSTOPERATİVE PAIN AFTER LAPAROSCOPIC HYSTERECTOMY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, Medical Doctor, associate professor, Erzincan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MUGLA-6
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Prior to starting surgery after general anesthesia, the 10 mL of normal saline was performed by the primary surgeon. The syringe was injected with 5 mL on each side into the cervical stroma at 3 and 9 o'clock with a depth of 2 to 3 cm.
  Interventions: Procedure: Para-cervical block
- Study (Experimental): Prior to starting surgery after general anesthesia, thE 10 mL of 0.5% bupivacaine with epinephrine was performed by the primary surgeon. The syringe was injected with 5 mL on each side into the cervical stroma at 3 and 9 o'clock with a depth of 2 to 3 cm.
  Interventions: Procedure: Para-cervical block

INTERVENTIONS:
Procedure: Para-cervical block — Block of inferior hypogastric plexus with local anesthetic

SUMMARY:
Total hysterectomy is one of the most common surgical procedure in gynecology. The laparoscopic route for the performance of hysterectomies are on the rise [1]. The laparoscopic hysterectomy (TLH) procedure has several advantages over open surgery such as better cosmetic outcomes, faster recovery earlier return to normal activities and work [1-3]. Nonetheless, postoperative pain (PP) remains an issue that scuppers these advantages [1-3].

The incidence of PP after TLH has been reported to vary from 35% to 63% [4,5]. The origin of PP after laparoscopy is multifactorial and complex such as perioperative predicaments, including pneumoperitoneum, stretching of the intraabdominal cavity, the blood left in the abdomen, and dissection of the pelvic region [6-7]. A randomized controlled trial has demonstrated that there may be more intense pain and greater analgesia requirements in the immediate postoperative period after laparoscopic surgery than after laparotomy [8]. Further inquiry to intercept the advancement and decrease the severity of PP is prominent to further improve TLH.

Women undergoing TLH experience two different pain characteristics including incisional pain and visceral pain in the first hour after the operation [6]. These pains were most intense 30 min after TLH, gradually decreasing thereafter for postoperative 72 hr [6]. High levels of acute postoperative pain (APP) are pertain with an increment risk of chronic postsurgical pain so control of these acute pains in the urgent postoperative period is vital for faster amelioration.

Many attempts have been tried to control APP after THL, such as transverse abdominal plane blocks, superior hypogastric plexus block, local anesthetic injection to the port side, and reduced port caliber [9-12]. Para-cervical bloc (PCB) is believed to block the Frankenhouser nerve plexus that supplies the visceral sensory fibers to the uterus, cervix, and top of the vagina. Only two randomized studies have assessed the effect of PCB in THL, but several limitations such as the small sample size preclude drawing conclusions on PP after TLH. Thus, the primary goal of this randomized clinical trial was to investigate if PCB at the onset of surgery, as a part of enhanced recovery protocol, could improve patient recovery after THL.

ELIGIBILITY:
Inclusion Criteria:

-Patients undergoing total type A laparoscopic hysterectomy with or without additional surgery, such as salpingo-oophorectomy or salpingectomy

Exclusion Criteria:

* age < 18 years
* refusal to provide consent
* inability to understand the study questionnaire
* severe psychiatric or mental disorder
* American Society of Anesthesiologists (ASA) physical status classification > III
* history of regular narcotic use within 6 months of the surgery
* conversion to laparotomy
* operation time > 90 min
* Additional procedures

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-14 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) pain score | up to 1 hour after the procedure
  1 h postoperative visual analog scale (VAS) pain score

SECONDARY OUTCOMES:
the quality of postoperative recovery | Up to 24 hours after the procedure
  the quality of postoperative recovery according to the QoR-40 questionnaire scores at 24 hours after the surgical procedure
faces pain scale-revised score | up to 2,4,6,12 hours after the procedure
  Faces pain scale-revised score is an objective method of pain assessment in which facial expressions of the patient are assessed by the investigator

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Mugla Sıtkı Kocman University Education and Research Hospital, Muğla, Mentese
  - Kemal Güngördük, Menteşe, Muğla

REFERENCES:
- [Derived] Gungorduk K, Gulseren V, Tastan L, Ozdemir IA. Paracervical block before laparoscopic total hysterectomy: A randomized controlled trial. Taiwan J Obstet Gynecol. 2024 Mar;63(2):186-191. doi: 10.1016/j.tjog.2024.01.013. PMID 38485313